CLINICAL TRIAL: NCT02430207
Title: Study of Incidence of Pulmonary Embolism During Peroperative Period of Temporary Pacing Via Femoral Vein Versus Subclavian Vein in China
Brief Title: Incidence of Pulmonary Embolism During Temporary Pacing Via Femoral Versus Subclavian Vein
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Suqian People's Hospital (Unknown); The First People's Hospital of Kunshan (Other); Danyang People's Hospital of Jiangsu Province (Unknown); Jiangsu Taizhou People's Hospital (Other); Xinghua People's Hospital (Unknown); Jiangyin People's Hospital (Other); Qidong People's Hospital (Unknown); Wuxi No. 2 People's Hospital (Other); Nantong No. 1 People's Hospital (Unknown); Changzhou No.2 People's Hospital (Other); Xuzhou Medical University (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); Northern Jiangsu People's Hospital (Other); Rugao People's Hospital (Other); Xuzhou Central Hospital (Other)
Responsible Party: Principal Investigator, Minglong Chen, Vice Director of Division of Cardiology, The First Affiliated Hospital of Nanjing Medical University; Professor of Medicine, Nanjing Medical University, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSN201407
Record Dates: First submitted 2015-04-21; First posted 2015-04-30 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2015-04

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; Temporary Pacing; Femoral Vein; Subclavian Vein
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Femoral Vein (Experimental): patients receiving temporary pacing via femoral vein
  Interventions: Procedure: temporary pacing femoral vein
- Subclavian Vein (Experimental): patients receiving temporary pacing via subclavian vein
  Interventions: Procedure: temporary pacing subclavian vein

INTERVENTIONS:
Procedure: temporary pacing femoral vein — Temporary pacing via femoral or subclavian vein
  Arms: Femoral Vein
Procedure: temporary pacing subclavian vein
  Arms: Subclavian Vein

SUMMARY:
Temporary pacing via femoral vein is used widely in mainland China, because of its feasibility and simplicity. However, pulmonary embolism often occurred after the procedure. It is not known that whether there was any difference in incidence of pulmonary embolism between via different approaches. This randomized and multi-center study was designed to verify whether temporary pacing via subclavian vein has lower incidence than via femoral vein.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* There is indication for temporary pacing
* Patients agreed to participate in the clinical trial and sign a written informed consent

Exclusion Criteria:

* History of pulmonary embolism or deep vein thrombosis
* Devices existing in vein system
* Patients who could not receive randomization
* Severe coagulation disorder
* Severe liver, kidney dysfunction
* Mental diseases
* Pregnancy
* Patients investigators believed not suitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants suffering from pulmonary embolism | 12 hours to 7 days after extraction of temporary pacing leads

SECONDARY OUTCOMES:
Percentage of participants suffering from deep vein thrombosis | 12 hours to 7 days after extraction of temporary pacing leads

CONTACTS AND LOCATIONS:
Overall Officials: Minglong Chen, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University

REFERENCES:
- [Background] ZOLL PM. Resuscitation of the heart in ventricular standstill by external electric stimulation. N Engl J Med. 1952 Nov 13;247(20):768-71. doi: 10.1056/NEJM195211132472005. No abstract available. PMID 13002611
- [Background] Gammage MD. Temporary cardiac pacing. Heart. 2000 Jun;83(6):715-20. doi: 10.1136/heart.83.6.715. No abstract available. PMID 10814641
- [Background] FURMAN S, SCHWEDEL JB. An intracardiac pacemaker for Stokes-Adams seizures. N Engl J Med. 1959 Nov 5;261:943-8. doi: 10.1056/NEJM195911052611904. No abstract available. PMID 13825713
- [Background] Cheng TO. Percutaneous transfemoral venous cardiac pacing. A simple and practical method. Chest. 1971 Jul;60(1):73-8. doi: 10.1378/chest.60.1.73. No abstract available. PMID 5571275
- [Background] Weinstein J, Gnoj J, Mazzara JT, Ayres SM, Grace WJ. Temporary transvenous pacing via the percutaneous femoral vein approach. A prospective study of 100 cases. Am Heart J. 1973 May;85(5):695-705. doi: 10.1016/0002-8703(73)90178-6. No abstract available. PMID 4697639
- [Background] Pandian NG, Kosowsky BD, Gurewich V. Transfemoral temporary pacing and deep vein thrombosis. Am Heart J. 1980 Dec;100(6 Pt 1):847-51. doi: 10.1016/0002-8703(80)90065-4. PMID 7446387
- [Background] Nolewajka AJ, Goddard MD, Brown TC. Temporary transvenous pacing and femoral vein thrombosis. Circulation. 1980 Sep;62(3):646-50. doi: 10.1161/01.cir.62.3.646. PMID 7398027
- [Background] Lopez Ayerbe J, Villuendas Sabate R, Garcia Garcia C, Rodriguez Leor O, Gomez Perez M, Curos Abadal A, Serra Flores J, Larrousse E, Valle V. [Temporary pacemakers: current use and complications]. Rev Esp Cardiol. 2004 Nov;57(11):1045-52. Spanish. PMID 15544753
- [Background] Klatsky AL, Armstrong MA, Poggi J. Risk of pulmonary embolism and/or deep venous thrombosis in Asian-Americans. Am J Cardiol. 2000 Jun 1;85(11):1334-7. doi: 10.1016/s0002-9149(00)00766-9. PMID 10831950
- [Background] Torbicki A, Perrier A, Konstantinides S, Agnelli G, Galie N, Pruszczyk P, Bengel F, Brady AJ, Ferreira D, Janssens U, Klepetko W, Mayer E, Remy-Jardin M, Bassand JP; ESC Committee for Practice Guidelines (CPG). Guidelines on the diagnosis and management of acute pulmonary embolism: the Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). Eur Heart J. 2008 Sep;29(18):2276-315. doi: 10.1093/eurheartj/ehn310. Epub 2008 Aug 30. PMID 18757870